CLINICAL TRIAL: NCT00419887
Title: A Randomized, Double-Blind, Placebo-Controlled, Time-Lagged, Parallel-Group, Ascending Single and Multiple Oral Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LAF237 in Chinese Healthy Subjects
Brief Title: Safety, Tolerability, Effect of Vildagliptin and How the Body Changes the Blood Level of Vildagliptin in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2109
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Safety, tolerability, pharmacokinetics, pharmacodynamics, LAF237, vildagliptin, Chinese, healthy volunteers
MeSH Terms: interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

INTERVENTIONS:
Drug: Vildagliptin (LAF237)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, effect of vildagliptin and how the body changes the blood level of vildagliptin of single and multiple oral doses of vildagliptin in healthy Chinese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy volunteers age 18 to 45 years of age included
* In good health as confirmed by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis on the screening and baseline evaluation
* All subjects must have both parents of Chinese origin and citizenship and must have been born in China.
* Body mass index (BMI) within the range of 19 to 24 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* Smokers
* Use of any prescription drugs within four (4) weeks prior dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within two (2) weeks prior to dosing. Paracetamol (or equivalent in China) is acceptable
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness within two weeks prior to dosing.
* A past personal or close family medical history of clinically significant cardiac abnormalities
* History of Acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease) Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis) Known hypersensitivity or severe adverse event to darifenacin or similar drugs Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize participation in the study Immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result. Drug or alcohol abuse within the 12 months prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2006-09

PRIMARY OUTCOMES:
Safety and tolerability of single dose of vildagliptin in healthy Chinese volunteers at four sequentially ascending dose levels
Safety and tolerability of repeated doses of vildagliptin in healthy Chinese volunteers at five sequentially ascending dose levels
Pharmacokinetics and pharmacodynamics of vildagliptin in healthy Chinese volunteers at five sequentially ascending dose levels

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamic relationship in healthy Chinese volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis, Beijing, China